CLINICAL TRIAL: NCT05228938
Title: Vaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) Salpingo-oophorectomy or Bilateral Salpingectomy Compared With Laparoscopic Approach. Prospective Study-A New Approach.
Brief Title: vNOTES Salpingo-oophorectomy or Bilateral Salpingectomy Compared With Laparoscopic.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment rate
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Meirav Braverman, Principal Investigator, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 114-21
Record Dates: First submitted 2021-11-02; First posted 2022-02-08 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Salpingectomy
Keywords: VNOTES; laparoscopic; Salpingo-oophorectomy; salpingectomy
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group: vNOTES (Experimental): Elective bilateral salpingectomy or Salpingo-oophorectomy by vaginal Natural Orifice Transluminal Endoscopic Surgery approach
  Interventions: Procedure: VNOTES
- Control group: Laparoscopic (Other): Elective bilateral salpingectomy or Salpingo-oophorectomy by conventional laparoscopy
  Interventions: Procedure: laparoscopic

INTERVENTIONS:
Procedure: VNOTES — vaginal Natural Orifice Transluminal Endoscopic Surgery approach for Elective bilateral salpingectomy or Salpingo-oophorectomy
  Arms: Study group: vNOTES
Procedure: laparoscopic — laparoscopic Surgery approach for Elective bilateral salpingectomy or Salpingo-oophorectomy
  Arms: Control group: Laparoscopic

SUMMARY:
Objective: To compare the vNOTES approach versus conventional laparoscopic approach used in elective Salpingo-oophorectomy surgery for benign disease or bilateral salpingectomy for sterilization.

Study design: Prospective cohort, randomized controlled trial.

Study population: Planned Salpingo-oophorectomy for benign disease or bilateral salpingectomy for sterilization.

Primary outcome - Adherence to planned surgical route, intra-operative parameters & complications, post-operative parameters & complications, rate of satisfaction.

DETAILED DESCRIPTION:
Objective: To compare the vNOTES approach versus conventional laparoscopic approach used in elective Salpingo-oophorectomy surgery for benign disease or bilateral salpingectomy for sterilization.

Study design: Prospective cohort, randomized controlled trial.

Study population: women aged over 18 who are planned to elective Salpingo-oophorectomy for benign disease or bilateral salpingectomy for sterilization.

Primary outcome - Removal of the ovaries and/or fallopian tubes according to the allocated technique, without conversion.

Secondary outcome - Duration of the surgical procedure, Duration of hospital admission (after surgery), The need for analgesics, and pain Numerical Rating Scale score , Post operation infection (up to 4 weeks from surgery), Need for medical examination/treatment or appearance of surgical complication up to 4 weeks form surgery (using Clavin Dindo Class), Bleeding assessment during surgery, Dyspareunia assessment - up to 3 months from surgery, Patient satisfaction from the surgical procedure will be measured with Patient Global Impression of Improvement (PGI-I).

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 18 and 80 years.
2. women who seek for definitive surgical sterilisation.
3. women who planed for Elective bilateral salpingectomy or Salpingo-oophorectomy for a non-malignant indication

Exclusion Criteria:

1. history of rectal surgery.
2. rectovaginal endometriosis
3. suspected malignancy
4. History of pelvic inflammatory disease.
5. active lower genital tract infection.
6. Virgo women
7. pregnancy
8. Failure to provide written informed consent prior to surgery

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-05-29 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Successful removal of the fallopian tubes or adnexa without a need to convert to another technique. | Intraoperative
  Number of Participants With Removal of the ovaries and/or fallopian tubes according to the allocated technique.

SECONDARY OUTCOMES:
Duration of surgical intervention | Intraoperative
  (Between incision and closure) in minutes
Duration of hospital admission after surgical intervention | from time of admission up to time of discharge from hospital
  Between surgery and time of discharge - in days
Bleeding assessment during surgical intervention | Intraoperative
  Estimation by the major surgeon of the quantity of bleeding during surgery - in ml The amount of blood in the vacuum container in the end of the surgery
Post operation infection | detected during the first six weeks of surgery
  Postoperative infection defined by lower abdominal pain with fever > 38°C and positive clinical signs or laboratory findings, detected during the first six weeks of surgery, as a dichotomous outcome
Postoperative pain scores | During the first seven days after the surgical intervention
  Postoperative pain scores, measured using a Visual Analogue Scale (VAS) twice daily (morning and evening) from day 1 till 7 selfreported by the participating women. VAS scores from 0 to 10 with 0 = no pain and 10= worst pain ever imaginable.
The use of analgetic drugs for postoperative pain | During the first week after the surgical intervention
  Postoperative pain defined by the total amount of analgesics used, as a continuous outcome.
Intra- Operative Complications | Intraoperative
  Intra- operative complications according to the Clavien- Dindo classification detected during the first six weeks of surgery, as a dichotomous outcome
Postoperative Complications | During the first six weeks after the surgical intervention
  Postoperative complications detected during the first 6 weeks of surgery, as a dichotomous outcome
Vaginal Pain During Sexual Intercourse at Three Months | At 3 months after the surgical intervention
  Incidence of vaginal dyspareunia recorded by the participants at 3 months by self-reporting using a simple questionnaire, as a dichotomous outcome
Patient satisfaction from the surgical procedure | At 3 months after the surgical intervention
  rate of satisfacation estimated with Patient Global Impression of Improvement questionnaire (PGI-I) . (score 1-7)
Hospital Readmission | During the first six weeks after the surgical intervention
  The number of women readmitted to hospital within six weeks following surgery, as a dichotomous outcome.

CONTACTS AND LOCATIONS:
Overall Officials: meirav braverman, MD, Principal Investigator — haemek medical center; Sivan Witzman, Study Director — haemek medical center; eyal rom, MD, Principal Investigator — haemek medical center
Locations (1):
- Haemek Medical Center, Afula, Israel